CLINICAL TRIAL: NCT05964959
Title: Dry Mouth in Patients With a Life-limiting Condition or Frailty: the Effect of a Nurse-led Patient Education Program
Brief Title: A Mouth Education Program for Dry Mouth
Acronym: MEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Yvette M. van der Linden, Prof. dr., Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL08440012010001
Record Dates: First submitted 2023-06-30; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Xerostomia; End of Life; Frailty; Dry Mouth
Keywords: Palliative Care; Educational Program; Oral Health
MeSH Terms: conditions — Xerostomia; Death; Frailty

STUDY DESIGN:
Intervention Model Description: A cluster-based intervention study in 6 hospitals and 6 nursing homes (n=228), followed by a mixed-methods study and cost-effective analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In the intervention group, the nurse and participant will be using the Mouth Education Program (MEP) to discuss causes, consequences and interventions for dry mouth in a structured manner, ultimately leading to an appropriate, individual treatment plan.
  The MEP is based on current clinical, national palliative care guidelines on dry mouth care.
  Interventions: Other: Mouth Educational Program
- Control (Active Comparator): The control group will receive care as usual, provided by their trusted, treating clinicians and care teams. Questionnaires will be administered by researchers.
  Interventions: Other: Care as Usual

INTERVENTIONS:
Other: Mouth Educational Program — The Mouth Educational Program is a nurse-led patient education program for dry mouth in patients with a life-limiting condition or frailty.
  Arms: Intervention
Other: Care as Usual — Care as usual is defined as the standard dry mouth care as provided by participants' own treating physicians.
  Arms: Control

SUMMARY:
The goal of this cluster based intervention trial is to evaluate the effect of a nurse-led patient education program on dry mouth in patients with a life-limiting condition or frailty.

The Mouth Educational Program (MEP) is a nurse-led patient education program, in which trained nurses use current clinical, palliative dry mouth guidelines in a structured manner to discuss causes, consequences and interventions with the patients and to create an appropriate treatment plan. This intervention will be compared to a control group receiving care as usual.

Therefore, the main question it aims to answer is:

Does a nurse-led patient education program reduce dry mouth complaints in patients with a life-limiting condition or frailty?

Participants will be asked to answer questionnaires and, when part of the intervention group, partake in the Mouth Educational Program (MEP).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* life-limiting condition or frailty (definition from Kwaliteitskader Palliatieve Zorg Nederland (IKNL/Palliactief, 2017)),
* experience the complaint dry mouth ≥ 5 on an 11 point numerical rating scale (ranging from 0=no dry mouth to 10=worst dry mouth ever);
* fulfil the Surprise Question (SQ): 'Would I be surprised if my patient dies within the year? (no)

Exclusion Criteria:

* life expectancy less than 4 weeks;
* previous medical history of radiotherapy to the salivary glands or Sjogren's syndrome;
* a cognitive inability to understand and participate in an educational program (assessed by a member of the regular care team, either doctor or nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage responders at week 4, as compared to baseline in both groups | Baseline to Week 4
  A responder is defined as a participant with a clinically relevant response, i.e. at least a 2-point reduction on the 11-point Numeric Rating Score (NRS) for dry mouth severity. The NRS ranges from 0=no dry mouth to 10=worst possible dry mouth.

SECONDARY OUTCOMES:
Change in mean Numeric Rating Score (NRS) for dry mouth severity upon MEP participation, as compared to the control group | Baseline to week 2, 4, 8 and 12
  Change in mean NRS dry mouth scores in the MEP group at all time-points when compared to the control group. The NRS ranges from 0=no dry mouth to 10=worst possible dry mouth.
Percentage responders at week 8 and 12, as compared to baseline in both groups | Baseline to Week 8 and 12
  A responder is defined as a participant with a clinically relevant response, i.e. at least a 2-point reduction on the 11-point Numeric Rating Score (NRS) for dry mouth severity. The NRS ranges from 0=no dry mouth to 10=worst possible dry mouth.
Change in dry mouth symptoms upon MEP participation as compared to the control group | Baseline to week 2, 4, 8 and 12
  Dry mouth symptoms are measured by the summated Xerostomia Inventory-Dutch Version (sXI-D). The sXI-D contains 5 items adressing dry mouth in general, dry mouth during eating, difficulty eating, difficulty swallowing and dry lips. Here, three items have been added: oral pain, difficulty speaking and change in taste. The sXI-D scale ranges from 0=never, 1=occassionally to 2=often.
Change in Oral Health-Related Quality of Life (OHRQoL) upon MEP participation, as compared to the control group | Week 4 to Week 8 and 12
  The OHRQoL is measured using the validated Dutch version of the Geriatric Oral Health Assessment Index (GOHAI-NL). The GOHAI-NL contains 12 items in three categories: phsyical function, psychosocial function and pain/discomfort, and uses a 5-point Likert scale ranging from 0=never to 5=often/always.
Change in clinical functioning upon MEP participation, as compared to the control group | Baseline to week 2, 4, 8 and 12
  Clinical functioning is examined by a patient-reported functional status (PRFS) scale. The PRFS was originally part of the validated Patient-Generated Subjective Global Assessment (PG-SGA) but has also been validated as a stand-alone measure. Activities and function are measured on a five-point scale, with the following definitions: 0= normal with no limitations, 1=not my normal self, but able to be up and about with fairly normal activities, 2=not feeling up to most things, but in bed or chair less than half of the day, 3=able to do little activity and spend most of the day in bed or chair, 4=bed ridden, rarely out of bed.
Change in Global Perceived Effect by participants upon MEP participation, as compared to the control group | Baseline to week 2, 4, 8 and 12
  GPE by participants is determined using a 7-point GPE scale. The GPE addresses perceived improvement of their condition, ranging from 1=very good, 2=good, 3=fairly good, 4=same as before, 5=fairly bad, 6=bad, 7=very bad.
Change in Health Related Quality of Life (HRQoL) upon MEP participation, as compared to the control group | Baseline to week 2, 4, 8 and 12
  The HRQoL is assessed using the EuroQoL five-demensional five-level questionnaire (EQ-5D-5L). The EQ-4D-4L contains five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 answer categories (levels): 0=no problems, 1=some problems, 2=moderate problems, 3=severe problems, and 4=extreme problems/unable to.

OTHER OUTCOMES:
Current clinical practices in dry mouth care as reported by health care professionals in both the control and intervention group (nurses and medical doctors) | At baseline and upon full study completion per study site (expected after an average of 1 year)
  Current clinical practices for dry mouth care as reported by health care professionals are examined by a self-developed questionnaire, including questions (open-ended and multiple choice) on work experience and education and on all aspects of clinical practice for dry mouth care (such as initial identification of dry mouth symptoms, medical anamnesis, physical examination, interventions/treatment and monitoring, and use of guidelines). The questionnaire will be administered to all participating nurses in the intervention and control group, and supplemented by at least one medical doctor per study site.
Current clinical practices in dry mouth care as experienced by participants in the control group | Week 12
  Participants' experiences in the control group (receiving care as usual) with dry mouth care are examined by individual semi-structured interviews.
Barriers and facilitators of the MEP as perceived by nurses participating in the intervention group. | Upon study completion, after an average of 1 year
  Barriers and facilitators as perceived by nurses leading the MEP consultations are identified through a questionnaire, adapted from the validated Dutch Implementation of an Innovation questionnaire. This questionnaire includes personal, logistic, financial, educational and work environment barriers and facilitators.
Barriers, facilitators and overall applicability of the MEP as a means to structurally implement the existing guidelines as perceived by nurses participating in the intervention group. | Upon study completion, after an average of 1 year
  The barriers, facilitators and overall applicability of the MEP as perceived by the nurses leading the MEP consultations is further explored in focus groups.
Barriers and facilitators of the MEP as perceived by participants in the intervention group. | Upon study completion, after an average of 1 year
  Experiences with the MEP and received care, including barriers and facilitators, by participants in the intervention group are examined by individual semi-structured interviews.
Barriers and facilitators of the current guidelines for dry mouth care in the Netherlands as perceived by nurses in both the intervention and control group. | Upon study completion, after an average of 1 year
  Barriers and facilitators of the current guidelines are examined in focus groups with nurses from either arm.
Cost-effectiveness Analysis (CEA) of the MEP, as compared to the control group | Week 0, 4, 8 and 12.
  The CEA is based upon patient-reported medical costs as measured by the Institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ). It encompasses use of medical and paramedical treatments or services, in- and outpatient care and use of medication. Here, the questionnaire consists of three main questions asking for the frequency of contact with dental services, the frequency of contact with health care professionals across different disciplines and the purchase of dry mouth treatment products (e.g. medication and other aids) in the last four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette M van der Linden, Prof. dr., Principal Investigator — Leiden University Medical Centre
Locations (1):
- Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The full IPD sharing plan or data sharing agreement can be provided upon request, but is based on the FAIR data sharing principles.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Only after completion of the total study and after publication by the original researchers, will data be made available.
Access Criteria: Data will be made available upon reasonable request by other researchers and will be decided upon on a case by case basis by the original researchers. When shared, data will be solely anonymized.

REFERENCES:
- [Derived] van der Meulen AI, Neis EPJG, de Nijs EJM, Coenegracht BJEG, Stoppelenburg A, van den Beuken-van Everdingen MHJ, van der Linden YM. Dry mouth in patients with a life-limiting condition or frailty: a study protocol for two intervention studies and a nested qualitative sub-study (the Dry mOuth Project, DROP). BMC Palliat Care. 2023 Aug 23;22(1):120. doi: 10.1186/s12904-023-01242-0. PMID 37612654